CLINICAL TRIAL: NCT02272946
Title: Effect of IL--1β Inhibition on Inflammation and Cardiovascular Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Priscilla Hsue, MD (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Priscilla Hsue, MD, Professor of Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Canakinumab
Record Dates: First submitted 2014-10-13; First posted 2014-10-23 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: HIV; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Arm (Other): In Stage 1: all 10 subjects will receive 150 mg Canakinumab subcutaneous injection. This will be a preliminary safety study (before Stage II).
  Interventions: Drug: Canakinumab
- Canakinumab (Experimental): In Stage II: About 67 subjects will receive 150mg Canakinumab subcutaneous injection.
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): In Stage II: About 33 subjects will receive 150mg placebo subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — 150mg Canakinumab received subcutaneously
  Other Names: IL--1β
  Arms: Canakinumab; Safety Arm
Drug: Placebo — 150mg Placebo received subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of IL-1β inhibition on safety, measures of systemic and vascular inflammation and endothelial function (all indicators of cardiovascular risk) in treated and suppressed HIV infected individuals This study will assess the safety and effects of canakinumab on endothelial function (assessed by flow-mediated vasodilation [FMD] of the brachial artery), vascular inflammation (assessed by FDG-PET/CT scanning), key inflammatory markers of cardiovascular disease (CVD) risk (high-sensitivity C-reactive protein [hsCRP]), interleukin-6 (IL-6), soluble CD163 (sCD163), D-dimer, T-cell and monocyte activation in the blood, and size of the HIV reservoir. 10 individuals will receive a single dose of 150mg canakinumab with follow-up for 12 weeks. In the second part of the study, 100 participants will be randomized (2:1 - canakinumab to placebo) and will be followed by for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection,
2. Age ≥ 40 years < 60 years
3. On continuous ART for at least 12 months with no change in regimen in 12 weeks prior to study entry
4. CD4+ T cell count ≥ 400 cells/mm3
5. HIV RNA level below the standard limit of quantification for 52 weeks prior to entry
6. High risk for CAD as defined by either documented CVD (including prior MI) or diabetes mellitus or 1 CVD risk factor (current smoking, hypertension, dyslipidemia, or hsCRP≥2mg/L.)
7. Individuals on stable doses of lipid lowering therapy and/or anti-hypertensive medication will be allowed in the study.
8. Appropriate documentation from medical records of prior receipt of pneumococcal vaccinations

Exclusion Criteria:

1. Women of childbearing potential or pregnant/nursing women
2. CABG surgery in the past 3 years
3. Class IV heart failure
4. Uncontrolled HTN
5. History of tuberculosis or latent TB that is not treated
6. Nephrotic syndrome or eGFR< 30 ml/min/1.73m2
7. Active hepatic disease or active/chronic hepatitis B or C
8. Any prior malignancy including KS
9. Serious illness requiring hospitalization or active infection requiring antibiotics within 90 days
10. Requirement for live active vaccination 3 months prior to, during, and 3 months after study
11. Concurrent immune modulating therapy
12. Diabetes Mellitus
13. History of multiple imaging studies associated with radiation exposure
14. Neutropenia defined as ANC<1500/mm
15. Triglycerides>400 mg/dL
16. History of hypersensitivity to study drug
17. History of EBV-related lymphoproliferative disorders
18. Active or untreated latent TB infection

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09; Primary Completion 2021-02 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Kentoffio K, Temu TM, Shakil SS, Zanni MV, Longenecker CT. Cardiovascular disease risk in women living with HIV. Curr Opin HIV AIDS. 2022 Sep 1;17(5):270-278. doi: 10.1097/COH.0000000000000756. Epub 2022 Jul 5. PMID 35938460
- Available data/document: Clinical Study Report — https://drive.google.com/open?id=1n47RTe3nB2_aPQTCXkkTfYodX-gnWKLE — The link above shows the current enrollment table of the Canakinumab study as of March 2, 2020.
- Available data/document: IL-1B inhibition [by way of Canakinumab] Reduces Atherosclerotic Inflammation in HIV Infection - Journal of the American College of Cardiology — https://linkinghub.elsevier.com/retrieve/pii/S0735-1097(18)38665-0 — The link above is the research publication written by Dr. Hsue (Primary Investigator) about how IL-1B inhibition [by way of Canakinumab] reduces atherosclerotic inflammation in the setting of HIV.

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Arm: In Stage 1: all 10 participants received 150 mg Canakinumab subcutaneous injection. This will be a preliminary safety study (before Stage II).
  Canakinumab: 150mg Canakinumab received subcutaneously
- Canakinumab: In Stage II: 25 participants received150mg Canakinumab subcutaneous injection.
  Canakinumab: 150mg Canakinumab received subcutaneously
- Placebo: In Stage II: 8 participants received 150mg placebo subcutaneous injection
  Placebo: 150mg Placebo received subcutaneously
Period: Overall Study
Arm/Group | Safety Arm | Canakinumab | Placebo
Started | 10 | 25 | 8
Completed | 10 | 25 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population are men or women who are at least 40 years, on stable anti-retroviral therapy and have documented cardiovascular disease or at risk for cardiovascular disease.
Groups:
- Canakinumab: In Stage II: 22 subjects will receive 150mg Canakinumab subcutaneous injection.
  Canakinumab: 150mg Canakinumab received subcutaneously
- Placebo: In Stage II: About 11 subjects will receive 150mg placebo subcutaneous injection
  Placebo: 150mg Placebo received subcutaneously
- Total: Total of all reporting groups
Arm/Group | Safety Arm | Canakinumab | Placebo | Total
Number analyzed (Participants) | 10 | 25 | 8 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 21 | 7 | 37
  >=65 years | 1 | 4 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 9 | 23 | 8 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 25 | 7 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 5 | 0 | 7
  White | 8 | 20 | 7 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Hypertension [Count of Participants; unit: Participants] | 9 | 10 | 2 | 21
Cardiovascular Disease [Count of Participants; unit: Participants] — Cardiovascular is defined as prior myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention, or luminal stenosis of at least 50% in at least one coronary artery.
  Participants | 3 | 2 | 1 | 6
Diabetes [Count of Participants; unit: Participants] | 3 | 2 | 3 | 8
Dyslipidemia on Statin Therapy [Count of Participants; unit: Participants] | 8 | 17 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in CD4 Count From Baseline to Follow-up
Description: Change in CD4 count from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log cells per mm^3
Groups:
- Canakinumab: In Stage II: 25 participants received 150mg Canakinumab subcutaneous injection.
  Canakinumab: 150mg Canakinumab received subcutaneously
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log cells per mm^3
  Week 4 | -0.085 [-0.170 to 0.008] | -0.024 [-0.106 to 0.065] | -0.020 [-0.149 to 0.129]
  Week 8 | -0.090 [-0.174 to 0.003] | 0.004 [-0.084 to 0.100] | -0.015 [-0.145 to 0.134]
  Week 12 | -0.049 [-0.139 to 0.050] | -0.111 [-0.186 to -0.029] | -0.070 [-0.192 to 0.072]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | -0.105 [-0.182 to -0.020] | -0.009 [-0.140 to 0.142]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | -0.142 [-0.220 to -0.057] | -0.012 [-0.147 to 0.145]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | -0.109 [-0.189 to -0.020] | -0.164 [-0.278 to -0.032]

2. Primary Outcome: Change in CD8 Count From Baseline to Follow-up
Description: Change in CD8 count from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log cells per mm^3
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log cells per mm^3
  Week 4 | -0.101 [-0.257 to 0.088] | -0.039 [-0.125 to 0.050] | 0.006 [-0.133 to 0.168]
  Week 8 | -0.103 [-0.259 to 0.086] | -0.069 [-0.154 to 0.030] | -0.040 [-0.173 to 0.115]
  Week 12 | -0.166 [-0.313 to 0.014] | -0.192 [-0.264 to -0.110] | -0.111 [-0.234 to -0.032]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | -0.202 [-0.274 to -0.120] | -0.098 [-0.223 to 0.047]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | -0.159 [-0.239 to -0.070] | -0.020 [-0.160 to 0.145]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | -0.171 [-0.250 to -0.080] | -0.198 [-0.313 to -0.063]

3. Primary Outcome: Change in Absolute Neutrophil Count From Baseline to Follow-up
Description: Change in absolute neutrophil count from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log unit (k) per uL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log unit (k) per uL
  Week 4 | -0.157 [-0.329 to 0.060] | -0.149 [-0.244 to -0.040] | -0.048 [-0.215 to 0.155]
  Week 8 | -0.137 [-0.314 to 0.084] | -0.015 [-0.130 to 0.120] | 0.044 [-0.139 to 0.266]
  Week 12 | -0.065 [-0.262 to 0.184] | -0.088 [-0.192 to 0.030] | 0.046 [-0.137 to 0.269]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | -0.110 [-0.213 to 0.010] | 0.053 [-0.131 to 0.278]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | -0.123 [-0.229 to 0.000] | 0.028 [-0.159 to 0.256]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | 0.056 [-0.072 to 0.200] | 0.201 [-0.017 to 0.468]

4. Primary Outcome: Change in Platelet Count From Baseline to Follow-up
Description: Change in platelet count from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log unit (k) per uL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log unit (k) per uL
  Week 4 | -0.098 [-0.168 to -0.022] | -0.079 [-0.131 to -0.020] | 0.026 [-0.066 to 0.127]
  Week 8 | -0.029 [-0.104 to 0.053] | -0.032 [-0.089 to 0.030] | 0.007 [-0.083 to 0.107]
  Week 12 | -0.014 [-0.093 to 0.072] | -0.020 [-0.076 to 0.040] | 0.014 [-0.077 to 0.115]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | 0.015 [-0.044 to 0.080] | 0.028 [-0.065 to 0.129]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | 0.016 [-0.046 to 0.080] | 0.054 [-0.044 to 0.162]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | 0.045 [-0.018 to 0.110] | -0.016 [-0.107 to 0.085]

5. Primary Outcome: Change in Creatinine Count From Baseline to Follow-up
Description: Change in creatinine count from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log mg/dL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log mg/dL
  Week 4 | -0.017 [-0.047 to 0.013] | 0.032 [-0.011 to 0.076] | -0.011 [-0.076 to 0.059]
  Week 8 | -0.001 [-0.030 to 0.030] | 0.014 [-0.029 to 0.059] | -0.012 [-0.078 to 0.057]
  Week 12 | -0.001 [-0.032 to 0.031] | -0.030 [-0.070 to 0.013] | -0.037 [-0.103 to 0.034]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | -0.017 [-0.059 to 0.026] | -0.068 [-0.129 to -0.002]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | -0.004 [-0.048 to 0.043] | -0.008 [-0.076 to 0.065]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | 0.014 [-0.032 to 0.061] | -0.037 [-0.103 to 0.034]

6. Primary Outcome: Change in AST From Baseline to Follow-up
Description: Change in AST from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log AST U/L
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log AST U/L
  Week 4 | 0.032 [-0.046 to 0.116] | 0.025 [-0.078 to 0.138] | -0.103 [-0.122 to 0.235]
  Week 8 | -0.019 [-0.093 to 0.061] | 0.001 [-0.102 to 0.115] | 0.055 [-0.110 to 0.250]
  Week 12 | 0.019 [-0.060 to 0.105] | 0.080 [-0.029 to 0.202] | 0.070 [-0.103 to 0.277]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | 0.024 [-0.081 to 0.141] | 0.069 [-0.098 to 0.268]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | 0.031 [-0.080 to 0.155] | -0.040 [-0.196 to 0.146]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | 0.008 [-0.100 to 0.130] | 0.049 [-0.121 to 0.251]

7. Primary Outcome: Change in ALT From Baseline to Follow-up
Description: Change in ALT from baseline (entry) to follow-up at weeks 4, 8, 12, 18, 24, and 36.
Time Frame: weeks 4, 8, 12, 18, 24, and 36.
Population: Safety only includes 10 individuals enrolled who received open label canakinumab and followed up to week 12.
Measure: Median (Inter-Quartile Range); unit: log ALT U/L
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
log ALT U/L
  Week 4 | 0.100 [-0.134 to 0.398] | 0.079 [-0.034 to 0.206] | -0.024 [-0.185 to 0.168]
  Week 8 | -0.123 [-0.310 to 0.114] | 0.046 [-0.067 to 0.172] | 0.116 [-0.068 to 0.336]
  Week 12 | 0.098 [-0.142 to 0.406] | 0.111 [-0.007 to 0.243] | 0.087 [-0.098 to 0.311]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | 0.092 [-0.26 to 0.224] | 0.140 [-0.048 to 0.364]
  Week 24: number analyzed (Participants) | 0 | 25 | 8
  Week 24 |  | 0.038 [-0.080 to 0.170] | 0.052 [-0.127 to 0.268]
  Week 36: number analyzed (Participants) | 0 | 25 | 8
  Week 36 |  | 0.007 [-0.107 to 0.136] | 0.205 [0.000 to 0.453]

8. Secondary Outcome: Flow-Mediated Dilation (FMD)
Description: Brachial artery FMD is calculated as the percentage increase in brachial artery diameter with hyperemia (an increase in the quantity of blood flow to a body part) induced relative to the resting brachial artery diameter. Percentage of brachial artery diameter is measured as FMD diameter/basal diameter
Time Frame: Baseline and Week 12
Population: The safety arm is an open label study where brachial artery FMD was measured at baseline and week 8.
Measure: Mean (Inter-Quartile Range); unit: Percent change in artery diameter
Groups:
- Placebo: In Stage II: 8 participants received placebo subcutaneous injection
  Placebo: 150mg Placebo received subcutaneously
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
Percent change in artery diameter
  Baseline FMD at 45 Seconds | 3 [2 to 5] | 3 [2 to 4] | 3 [3 to 5]
  Baseline FMD at 60 Seconds | 4 [2 to 5] | 4 [2 to 6] | 4 [3 to 5]
  Baseline FMD at 75 Seconds | 4 [2 to 5] | 3 [2 to 5] | 3 [3 to 4]
  Baseline FMD at 90 Seconds | 2 [1 to 3] | 3 [2 to 4] | 2 [0 to 3]
  Week 12 FMD at 45 Seconds: number analyzed (Participants) | 0 | 25 | 8
  Week 12 FMD at 45 Seconds |  | 3 [2 to 4] | 4 [2 to 5]
  Week 12 FMD at 60 Seconds: number analyzed (Participants) | 0 | 25 | 8
  Week 12 FMD at 60 Seconds |  | 3 [2 to 6] | 4 [3 to 5]
  Week 12 FMD at 75 Seconds: number analyzed (Participants) | 0 | 25 | 8
  Week 12 FMD at 75 Seconds |  | 2 [2 to 6] | 4 [2 to 5]
  Week 12 FMD at 90 Seconds: number analyzed (Participants) | 0 | 25 | 8
  Week 12 FMD at 90 Seconds |  | 2 [1 to 4] | 3 [2 to 5]
  Week 8 FMD at 45 Seconds: number analyzed (Participants) | 10 | 0 | 0
  Week 8 FMD at 45 Seconds | 3 [2 to 3] |  |
  Week 8 FMD at 60 Seconds: number analyzed (Participants) | 10 | 0 | 0
  Week 8 FMD at 60 Seconds | 3 [2 to 4] |  |
  Week 8 FMD at 75 Seconds: number analyzed (Participants) | 10 | 0 | 0
  Week 8 FMD at 75 Seconds | 3 [2 to 4] |  |
  Week 8 FMD at 90 Seconds: number analyzed (Participants) | 10 | 0 | 0
  Week 8 FMD at 90 Seconds | 2 [1 to 4] |  |

9. Secondary Outcome: Arterial Inflammation Measured at Baseline and Follow-up at Week 12
Description: Change From Baseline in Arterial Fluorodeoxyglucose (FDG) Uptake Assessed by FDG-PET/CT and reported as target-to-background (TBR) ratio to measure of vascular inflammation
Time Frame: Baseline (entry) and Week 12
Measure: Mean (Standard Deviation); unit: target-to-background ratio
Groups:
- Placebo: In Stage II: 8 participants received placebo subcutaneous injection
  Placebo: Placebo received subcutaneously
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
target-to-background ratio
  Baseline (Entry) | 3.27 (0.57) | 3.18 (0.58) | 3.85 (1.14)
  Week 12 | 2.97 (0.64) | 3.21 (0.73) | 4.01 (0.78)

10. Secondary Outcome: D-Dimer
Description: D-Dimer will be assessed from baseline to weeks 4, 8, 12, and 18.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, and week 18
Population: The safety arm is an open label study with D-Dimer markers evaluated at baseline, week 4, and week 8.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 25 | 8
ng/mL
  Baseline | 548.3 [429.5 to 1040.1] | 2121.89 [1809.53 to 2970.82] | 1917.03 [1692.92 to 2092.69]
  Week 4 | 499.7 [373.1 to 1226] | 2042.96 [1905.96 to 3077.26] | 2080.01 [1388.74 to 2676.91]
  Week 8: number analyzed (Participants) | 10 | 0 | 0
  Week 8 | 562.4 [445.5 to 844.4] |  |
  Week 12: number analyzed (Participants) | 0 | 25 | 8
  Week 12 |  | 2126.05 [1766.84 to 2671.45] | 1894.52 [1548.59 to 2341.66]
  Week 18: number analyzed (Participants) | 0 | 25 | 8
  Week 18 |  | 1879.56 [1336.44 to 2551.52] | 1669.79 [1269.7 to 2402.89]

11. Secondary Outcome: Human Serum Amyloid A (SAA)
Description: SAA will be assessed from baseline to weeks 4, 12, and 18.
Time Frame: Baseline, 4 weeks, 12 weeks, and week 18
Population: The safety arm did not evaluate Human Serum Amyloid A
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 25 | 8
pg/mL
  Baseline |  | 479058.3 [263456 to 44598329] | 513209.75 [196985 to 842869.45]
  Week 4 |  | 310588.7 [240857.9 to 1323745] | 20045206 [2841774.5 to 37070079]
  Week 12 |  | 844889.8 [139007.15 to 4572776] | 1968440.05 [204694.55 to 36420571.5]
  Week 18 |  | 8838641 [2702749 to 19603171] | 615594.95 [147562.15 to 8188797]

12. Secondary Outcome: Tumor Necrosis Factor Alpha (TNFa)
Description: TNFa will be assessed from baseline to weeks 4, 12, and 18.
Time Frame: Baseline, 4 weeks, 12 weeks, and week 18
Population: The safety arm did not evaluate Tumor Necrosis Factor Alpha
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Safety Arm | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 25 | 8
pg/mL
  Baseline |  | 1.69 [1.3 to 2.04] | 1.24 [1.16 to 1.9]
  Week 4 |  | 1.47 [0.96 to 1.88] | 1.34 [1.13 to 2.19]
  Week 12 |  | 1.18 [0.9 to 1.44] | 1.4 [0.86 to 1.98]
  Week 18 |  | 1.16 [1.06 to 1.5] | 1.41 [1.01 to 1.63]

ADVERSE EVENTS:
Time Frame: 36 weeks
Groups:
- Safety Arm: In Stage 1: all 10 participants will receive 150 mg Canakinumab subcutaneous injection. This will be a preliminary safety study (before Stage II).
  Canakinumab: 150mg Canakinumab received subcutaneously
- Canakinumab: In Stage II: 25 participants will receive 150mg Canakinumab subcutaneous injection.
  Canakinumab: 150mg Canakinumab received subcutaneously
- Placebo: In Stage II: 8 participants will receive 150mg placebo subcutaneous injection
  Placebo: 150mg Placebo received subcutaneously
Arm/Group | Safety Arm | Canakinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/25 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/25 | 0/8
Other Adverse Events (participants affected / at risk) | 2/10 | 1/25 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Arm (N=10) | Canakinumab (N=25) | Placebo (N=8)
Kaposi Sarcoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Streptococcal Sepsis (Blood and lymphatic system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Arm (N=10) | Canakinumab (N=25) | Placebo (N=8)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02272946/Prot_SAP_000.pdf